CLINICAL TRIAL: NCT01517737
Title: Immune Cell Involvement in the Tissue Response to Metallosis in Patients With Failed Metal-on-metal Hip Replacements
Brief Title: Immunology of Failing Metal-on-Metal Hip Replacement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of East Anglia (Other)
Collaborators: Depuy, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011 Orth 04S (68-06-11); IIS2010015 (Other Grant/Funding Number: DePuy)
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Infection of Total Hip Joint Prosthesis; Implants

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — blood from all patients; joint fluid, soft tissue and bone on operated patients
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Metal-on-metal total hip replacement (MoM THR) has been targeted at younger patients with anticipated long-term survival since the bearing surfaces wear less than the traditional metal-on-plastic (MoP) replacements. However, the production of metal ions as a result of the wear is a concern because of the possible toxicity to cells. In Norwich England a number of different metal-on-metal implants have been trialed of which one, the Ultima TPS, has had very poor results. A total of 545 patients have had 652 MoM THRs with the Ultima TPS of whom more than 20% have now been revised. There is an ongoing MHRA program to screen for problems using MRI scans with a technique developed in Norwich. Investigations so far show massive corrosion in the implants with a catastrophic immune response causing death of cells. This may include death of bone leading to fracture. In a third of patients revised there has been pain but normal plain X-rays. In some patients without pain who have been screened there are abnormal changes on an MRI scan. We wish to investigate the immune cells in patients to find out why this has happened. The study will include patients coming for a new hip to act as a comparator, as well as those with a MoM THR and patients being revised with MoM THRs, and MoP THRs. We shall also investigate patients with other MoM THRs opportunistically.

DETAILED DESCRIPTION:
To characterize dendritic cell (DC) populations in MoM THR patients. Dendritic cells are cells that migrate from the circulating blood into tissues and mop up foreign material such as viruses with their abnormal surface makers (antigens)and metal debris, activating specialist white blood cells (such as T cells) that kill viruses and remove abnormal material.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone Ultima TPS THRs in Norwich
* Patients with a MoP THR under going revision.
* Patients undergoing primary hip replacement with osteoarthritis
* Patients with other MoM THRs undergoing revision

Exclusion Criteria:

* Patients undergoing primary THR with rheumatoid arthritis or other inflammatory arthritides, or secondary to infection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The Ultima TPS patients are all identified and regularly followed up. Other patients will be identified from planned operating lists and waiting lists. This will be carried out by the research team.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pinar Court, Principal Investigator — University of East Anglia
Locations (2):
- United Kingdom (2):
  - Norfolk and Norwich University Hospital NHS Trust, Norwich, Norfolk
  - Norfolk and Norwich University Hospital, Norwich, Norfolk